CLINICAL TRIAL: NCT00221455
Title: The Potential of Technology to Improve Chronic Disease Management and Quality of Care
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 51760; 51760
Record Dates: First submitted 2005-09-15; First posted 2005-09-22 (Estimated); Last update posted 2011-07-27 (Estimated); Status verified 2011-07

CONDITIONS: Diabetes Mellitus
Keywords: Diabetes Mellitus; Chronic disease management; Patient portal; Patient empowerment
MeSH Terms: conditions — Diabetes Mellitus; Patient Participation

INTERVENTIONS:
Behavioral: Patient diabetic self-management using the diabetic patient portal tools
Behavioral: A variety of educational interventions for non-adopters of the technology, and for non-compliant patients.

SUMMARY:
We seek to determine if patient data entry, data entered based alerts, and data review in a secure patient portal may provide a sustainable approach to improve diabetic outcomes in a cost effective manner. We plan to study the extent to which the portal can improve diabetic outcomes and quality of care. We recognize, however, that some patients will be more predisposed to adopting technology and some will be more predisposed to improving their compliance than others. Hence, we will also develop and test interventions that may improve adoption and compliance. The goals of the proposed study are: 1) to assess whether a web portal will improve care outcomes in diabetic patients; 2a) to describe the characteristics of patients whose health behavior improves over the study period; 2b) to describe the characteristics of patients who adopt the web portal-based disease management technology; 3) to develop and test targeted interventions to increase the adoption of the web portal and improve patient health behavior; and 4) to monitor the ongoing costs associated with the web portal and patient healthcare resource utilization, and to monitor the incremental costs of the interventions designed to improve utilization of the technology and patient compliance with their diabetic regimens.

DETAILED DESCRIPTION:
To date, limited research has been conducted to determine if health information technology (HIT) is effective in improving the outcomes for patients with chronic diseases. Research is required to determine if interventions facilitated by an institutional EMR platform can be implemented such that they support patients with chronic diseases to achieve improved outcomes in a cost effective fashion.

At the Cleveland Clinic Foundation (CCF) an ambulatory EMR has been implemented to foster patient safety and institutional best practice guidelines, to facilitate research, and to achieve efficiencies in practice management. Our EMR is the foundation of the CCF patient portal. One of the functions of the portal is to allow patients to enter specific data elements that become part of their permanent medical record. Diabetics can enter and review their home glucometer readings, and view alert messages based on their entries. The entries are transferred to the patient's primary care physician's EMR In-Basket for review.

We recognize that some patients will be more predisposed to technology adoption and some will be more health behavior compliant than others. Therefore, in addition to studying our portal's efficacy in positive diabetic behavior change, we will test if interventions can assist less predisposed and less compliant patients to become more compliant and more inclined to adopt the technology.

The goals of the proposed study are:

1) to assess whether a web portal will improve care outcomes in diabetic patients; 2a) to describe the characteristics of patients whose health behavior improves over the study period; 2b) to describe the characteristics of patients who adopt the web portal-based disease management technology; 3) to develop and test targeted interventions to increase the adoption of the web portal and improve patient health behavior; 4) to monitor the ongoing costs associated with the web portal and patient healthcare resource utilization, and to monitor the incremental costs of the interventions designed to improve utilization of the technology and patient compliance with their diabetic regimens.

ELIGIBILITY:
Inclusion Criteria: Diabetic patients 18 years of age or older with an established primary care physician at the Cleveland Clinic Foundation

Exclusion Criteria: An individual not meeting the inclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2004-09; Study Completion 2007-09 (Actual)

PRIMARY OUTCOMES:
Clinical Outcome Measures: HbA1c, LDL,and the presence or absence of clinically significant proteinuria.

SECONDARY OUTCOMES:
Technology Adoption will be measured by tracking the patient usage of the various portal features

CONTACTS AND LOCATIONS:
Overall Officials: Martin Harris, MD, MBA, Principal Investigator — The Cleveland Clinic; Holly D Miller, MD, MBA, Study Director — The Cleveland Clinic
Locations (1):
- The Cleveland Clinic Foundation, Cleveland, Ohio, United States

REFERENCES:
- [Background] Ajzen, I. (1991). The Theory of Planned Behavior. Organizational Behavior and Human Decision Processes, Vol. 50: 179-211.
- [Background] Avital, M., Vandenbosch, B., (2000) IT-Business Ownership: The Missing Link for IT-Driven Value, Administrative Sciences Association of Canada - 2000 Proceedings (Information Systems), Vol. 21(4): 116-125.
- [Background] Hogan P, Dall T, Nikolov P; American Diabetes Association. Economic costs of diabetes in the US in 2002. Diabetes Care. 2003 Mar;26(3):917-32. doi: 10.2337/diacare.26.3.917. PMID 12610059
- [Background] Beckles GL, Engelgau MM, Narayan KM, Herman WH, Aubert RE, Williamson DF. Population-based assessment of the level of care among adults with diabetes in the U.S. Diabetes Care. 1998 Sep;21(9):1432-8. doi: 10.2337/diacare.21.9.1432. PMID 9727887
- [Background] Biermann E, Dietrich W, Standl E. Telecare of diabetic patients with intensified insulin therapy. A randomized clinical trial. Stud Health Technol Inform. 2000;77:327-32. PMID 11187566
- [Background] Chang S., Ryoo S., Yu S., Ahn B., (1999) Development of an Internet-Based Home Monitoring System for Diabetes Mellitus, Proceeding of the 4th IEEE Malaysia International Conference on Communications and 4th IEEE Asia Pacific International Symposium on Consumer Electronics, Maleka, Malaysia, November 1999.
- [Background] Chase HP, Pearson JA, Wightman C, Roberts MD, Oderberg AD, Garg SK. Modem transmission of glucose values reduces the costs and need for clinic visits. Diabetes Care. 2003 May;26(5):1475-9. doi: 10.2337/diacare.26.5.1475. PMID 12716807
- [Background] Eisenberg JM. Ten lessons for evidence-based technology assessment. JAMA. 1999 Nov 17;282(19):1865-9. doi: 10.1001/jama.282.19.1865. No abstract available. PMID 10573279
- [Background] Fishbein M., Ajzen I., (1975) Belief, Attitude, Intention and Behavior: An Introduction to Theory and Research. Reading, MA: Addison-Wesley.
- [Background] Friedman RH, Stollerman JE, Mahoney DM, Rozenblyum L. The virtual visit: using telecommunications technology to take care of patients. J Am Med Inform Assoc. 1997 Nov-Dec;4(6):413-25. doi: 10.1136/jamia.1997.0040413. PMID 9391929
- [Background] Friedman RH, Stollerman J, Rozenblyum L, Belfer D, Selim A, Mahoney D, Steinbach S. A telecommunications system to manage patients with chronic disease. Stud Health Technol Inform. 1998;52 Pt 2:1330-4. PMID 10384677
- [Background] Gallagher, K., Vandenbosch, B., (2000) A Systemic View of Continual Change. Best Paper Proceedings of the Sixtieth Annual Meeting of the Academy of Management, August 2000.
- [Background] Hailey D, Roine R, Ohinmaa A. Systematic review of evidence for the benefits of telemedicine. J Telemed Telecare. 2002;8 Suppl 1:1-30. doi: 10.1258/1357633021937604. PMID 12020415
- [Background] Hersh WR, Helfand M, Wallace J, Kraemer D, Patterson P, Shapiro S, Greenlick M. Clinical outcomes resulting from telemedicine interventions: a systematic review. BMC Med Inform Decis Mak. 2001;1:5. doi: 10.1186/1472-6947-1-5. Epub 2001 Nov 26. PMID 11737882
- [Background] Kwon H., Cho J, Kim H., Song B., Ko S., Lee J., Kim S., Chang S., Kim H., Cha B., Lee K., Son H., Lee J., Lee W., Yoon K., (2004) Establishment of Blood Glucose Monitoring System Using the Internet, Diabetes Care, Vol. 27(2):478-83. Mease A, Whitlock W, Brown A, (2000) Telemedicine Improved Diabetic Management. Military Medicine, Vol. 165:279-284. Neubauer A., Priglinger S., Ehrt O., (2001) Electronic Versus Paper-Based Patient Records: a Cost-Benefit Analysis, Ophthalmologe, Vol. 11:1083-8. Norris S., Engelgau M., Narayan K., (2001) Effectiveness of Self-Managed Training in Type 2 Diabetes: A Systematic Review of Randomized Controlled Trials, Diabetes Care, Vol. 24/3.
- [Background] Olivarius NF, Beck-Nielsen H, Andreasen AH, Horder M, Pedersen PA. Randomised controlled trial of structured personal care of type 2 diabetes mellitus. BMJ. 2001 Oct 27;323(7319):970-5. doi: 10.1136/bmj.323.7319.970. PMID 11679387
- [Background] Piette JD, McPhee SJ, Weinberger M, Mah CA, Kraemer FB. Use of automated telephone disease management calls in an ethnically diverse sample of low-income patients with diabetes. Diabetes Care. 1999 Aug;22(8):1302-9. doi: 10.2337/diacare.22.8.1302. PMID 10480775
- [Background] Ralston JD, Revere D, Robins LS, Goldberg HI. Patients' experience with a diabetes support programme based on an interactive electronic medical record: qualitative study. BMJ. 2004 May 15;328(7449):1159. doi: 10.1136/bmj.328.7449.1159. PMID 15142919
- [Background] Renders CM, Valk GD, Franse LV, Schellevis FG, van Eijk JT, van der Wal G. Long-term effectiveness of a quality improvement program for patients with type 2 diabetes in general practice. Diabetes Care. 2001 Aug;24(8):1365-70. doi: 10.2337/diacare.24.8.1365. PMID 11473071
- [Background] Renders CM, Valk GD, Griffin SJ, Wagner EH, Eijk Van JT, Assendelft WJ. Interventions to improve the management of diabetes in primary care, outpatient, and community settings: a systematic review. Diabetes Care. 2001 Oct;24(10):1821-33. doi: 10.2337/diacare.24.10.1821. PMID 11574449
- [Background] Ross SE, Lin CT. The effects of promoting patient access to medical records: a review. J Am Med Inform Assoc. 2003 Mar-Apr;10(2):129-38. doi: 10.1197/jamia.m1147. PMID 12595402
- [Background] Schultze, U., Vandenbosch, B., (1998) Information Overload in a Groupware Environment: Now You See It, Now You Don't, Journal of Organizational Computing and Electronic Commerce, Vol. 8/2: 127-148.
- [Background] Shiffman RN, Liaw Y, Brandt CA, Corb GJ. Computer-based guideline implementation systems: a systematic review of functionality and effectiveness. J Am Med Inform Assoc. 1999 Mar-Apr;6(2):104-14. doi: 10.1136/jamia.1999.0060104. PMID 10094063
- [Background] Taylor S., Todd P., (1995). Understanding Information Technology Usage: A Test of Competing Models. Information Systems Research, Vol. 6(2), 144-176.
- [Background] Tierney WM, Miller ME, Overhage JM, McDonald CJ. Physician inpatient order writing on microcomputer workstations. Effects on resource utilization. JAMA. 1993 Jan 20;269(3):379-83. PMID 8418345
- [Background] Vandenbosch, B., (1995) Healthcare Data Exchange Corporation, In N. Lorenzi, R.T. Riley, M.J. Ball,& J.V. Douglas (Eds.), Transforming Health Care through Information: Case Studies, New York: Springer-Verlag, 337-350.
- [Background] Vandenbosch, B., (1995) What Makes an ESS Successful: Links Between Types of Use and Perceptions of Competitiveness, Administrative Sciences Association of Canada - 1995 Proceedings (Information Systems), Vol. 16/4: 97-106.
- [Background] Venkatesh, V. (2000) Determinants of Perceived Ease of Use: Integrating Control, Intrinsic Motivation and Emotion into the Technology Acceptance Model. Information Systems Research, Vol. 11(4) 342-365.
- [Background] Wagner EH, Grothaus LC, Sandhu N, Galvin MS, McGregor M, Artz K, Coleman EA. Chronic care clinics for diabetes in primary care: a system-wide randomized trial. Diabetes Care. 2001 Apr;24(4):695-700. doi: 10.2337/diacare.24.4.695. PMID 11315833
- [Background] Wang SJ, Middleton B, Prosser LA, Bardon CG, Spurr CD, Carchidi PJ, Kittler AF, Goldszer RC, Fairchild DG, Sussman AJ, Kuperman GJ, Bates DW. A cost-benefit analysis of electronic medical records in primary care. Am J Med. 2003 Apr 1;114(5):397-403. doi: 10.1016/s0002-9343(03)00057-3. PMID 12714130
- [Background] Whitten PS, Mair FS, Haycox A, May CR, Williams TL, Hellmich S. Systematic review of cost effectiveness studies of telemedicine interventions. BMJ. 2002 Jun 15;324(7351):1434-7. doi: 10.1136/bmj.324.7351.1434. PMID 12065269
- [Background] Wickramasinghe, N., Levitan, N., Vandenbosch, B., (1998) University Hospitals Automation, Prentice Hall Case Series in M.I.S.
- [Background] Yang, H., Vandenbosch, B., (1998) Visibility as the Basis of a Framework for Identifying Strategic Information Systems, Journal of Information Technology Management, Vol. 9/2, 31-42.
- See also: Patient portal log in page — https://mychart.clevelandclinic.org/default.asp